CLINICAL TRIAL: NCT00325455
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Efficacy, Safety, and Tolerability of MK-0859 in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia
Brief Title: MK0859 Dose-Ranging Study (0859-003)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-003; 2006_006
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Hypercholesterolemia; Mixed Hyperlipemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type V | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0859

SUMMARY:
To assess the cholesterol changing effects of MK0859 in patients with primary hypercholesterolemia or mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be men and women of non-child bearing potential, 18 through 75 years of age diagnosed with high cholesterol

Exclusion Criteria:

* Patients with CHD or CHD-equivalent disease (except diabetes)
* Diabetics on statins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess the cholesterol changing effects of MK0859

SECONDARY OUTCOMES:
Acceptable safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Dansky HM, Bloomfield D, Gibbons P, Liu S, Sisk CM, Tribble D, McKenney JM, Littlejohn TW 3rd, Mitchel Y. Efficacy and safety after cessation of treatment with the cholesteryl ester transfer protein inhibitor anacetrapib (MK-0859) in patients with primary hypercholesterolemia or mixed hyperlipidemia. Am Heart J. 2011 Oct;162(4):708-16. doi: 10.1016/j.ahj.2011.07.010. Epub 2011 Sep 1. PMID 21982664
- [Derived] Krauss RM, Pinto CA, Liu Y, Johnson-Levonas AO, Dansky HM. Changes in LDL particle concentrations after treatment with the cholesteryl ester transfer protein inhibitor anacetrapib alone or in combination with atorvastatin. J Clin Lipidol. 2015 Jan-Feb;9(1):93-102. doi: 10.1016/j.jacl.2014.09.013. Epub 2014 Oct 13. PMID 25670366